CLINICAL TRIAL: NCT04944875
Title: Effects of Music and Maternal Voice on Sedation Depth and Sedative Use During Pediatric
Brief Title: Effects of Music and Maternal Voice on Sedation Depth and Sedative Use During Pediatric Magnetic Resonance Imaging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem ÖZ GERGİN, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019/266
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Solid Tumor; Pediatric Brain Tumor; Pediatric Cancer
Keywords: Magnetic Resonance; sedation; maternal voice; sedative effects
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I; group headphone (Active Comparator): In the first group of the patients in the isolation group wear the headphones but do not listen to music during the procedure. Then patients were sedated by midazolam and propofol.
  Interventions: Procedure: Group headphone
- Group II; group music (Active Comparator): In the second group of the patients wear the headphones and listen to Vivaldi's The Four Seasons violin concertos by sound isolating headphones during the procedure.
  Then patients were sedated by midazolam and propofol.
  Interventions: Procedure: Group music
- Group III; group maternal voice (Active Comparator): In the third group of the patients wear the headphones and listen the maternal voice during the procedure.Then patients were sedated by midazolam and propofol.
  Interventions: Procedure: Group maternal voice

INTERVENTIONS:
Procedure: Group headphone — The patients in the first group wore the headphones but did not listen the music or maternal voice. The standard sedation method was applied to all patients.
  Arms: Group I; group headphone
Procedure: Group music — The patients in the second group listened to classical music (Vivaldi's The Four Seasons violin concertos) by sound- isolating headphones through the procedure.The standard sedation method was applied to all patients.
  Arms: Group II; group music
Procedure: Group maternal voice — The patients in the third group listened to maternal voice by sound- isolating headphones through the procedure.The standard sedation method was applied to all patients.
  Arms: Group III; group maternal voice

SUMMARY:
To evaluate the effects of music and maternal voice in children on sedation depth and sedative use during pediatric magnetic resonance imaging.

DETAILED DESCRIPTION:
When the patients and their parents arrived in the magnetic resonance unıt about 30 minutes before the procedure, the anesthetist is obtained a medical history and carried out a physical examination and clinical assesment.

Patients were categorized into 3 groups: music, maternal voice and isolation. During the procedures,the patients in the music group listened to Vivaldi's The Four Seasons violin concertos by sound isolating headphones, whereas the patients in the isolation group wore the headphones but did not listen to music.

All patients were sedated by midazolam and propofol. During the procedure, an additional propofol was administered as required

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I-II

Exclusion Criteria:

* Patients with hearing impairment, distorted ear anatomy, recent organ or system deficiency, severe pulmonary and/or cardiovascular problems, intolerance to propofol, airway ab-normalities, or known psychiatric or mental problems were ex-cluded from the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
amount of propofol dose used in sedation | during the MRI procedure
  The total propofol dosage were recorded in during procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Oz Gergin, Principal Investigator — TC Erciyes University
Locations (1):
- Özlem Öz Gergin, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 24 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.

REFERENCES:
- [Background] Starkey E, Sammons HM. Sedation for radiological imaging. Arch Dis Child Educ Pract Ed. 2011 Jun;96(3):101-6. doi: 10.1136/adc.2008.153072. Epub 2010 Jul 30. No abstract available. PMID 20675522
- [Background] Ahmad R, Hu HH, Krishnamurthy R, Krishnamurthy R. Reducing sedation for pediatric body MRI using accelerated and abbreviated imaging protocols. Pediatr Radiol. 2018 Jan;48(1):37-49. doi: 10.1007/s00247-017-3987-6. Epub 2018 Jan 1. PMID 29292482